CLINICAL TRIAL: NCT02488239
Title: Optimizing Pacing Therapy by Using Multi-Programmable Pulse Generators for Cardiac Resynchronization Pacing (CRT-P)
Acronym: Rally CRT-P
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: Rally-CRT-P-02-2015
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-03

CONDITIONS: Post Market Surveillance Study Following Clinical Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT-P indicated patients: Planned to be implanted with a 3-lead CRT-P system and connected to the remote data collection through the Latitude® system
  Interventions: Device: CRT-P indicated patients

INTERVENTIONS:
Device: CRT-P indicated patients — Patients who are indicated for a CRT-P device are planned to be implanted with a CRT-P device
  Other Names: Pacemaker implant

SUMMARY:
The objective of this Post Market Clinical Follow-up (PMCF) is to collect data on the performance of the Ingenio 2 CRT-P devices and to document that device-related events, device malfunctions or device deficiencies (DDs) do not increase safety risks in Ingenio 2 CRT-P devices (CRT-Ps), both in general and specific to the new features and hardware of the devices.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center, single group, post market clinical study The devices are fully commercially available and all subjects are planned to receive a CRT-P implant as part of their standard of care (SOC). The assignment of the specific Ingenio 2 device is physician's choice and will consider leads currently in place from previous devices and planned new leads (e.g., Acuity X4 and/or other LV leads).

Enrollment and Consenting Clinic Visit (≤ 30 days prior to implant procedure) (required)

* Implant Procedure (Day 0; all future follow ups based on this date) (required)
* Pre-Discharge Clinic Visit (after pocket closure and wound coverage 0-5 days post-implant procedure) (required)
* 1 month post-implant Clinic Visit (30 ± 15 days) (required)
* 3 month post-implant Clinic Visit (91 ± 21 days) (required)
* Latitude-based Close-out (91 - 120 days months post last enrollment) (reporting only required)
* Unscheduled clinic follow-up (any clinic visit between pre-discharge and 3 month follow up which is in addition to the 1 month follow up; per center SOC or subject needs; event reporting only)
* Re-implant/Revision (as needed)
* During the trial unanticipated serious adverse device effects (USADEs), serious adverse device effects (SADEs), adverse device effects (ADEs), DDs, all serious adverse events (SAEs), deaths, and changes in the device system must be reported (enrollment to Closeout).

Study Duration Enrollment is expected to take 12 months. The study will be considered complete (primary endpoint completion) after all subjects have completed the Latitude based close-out 3-4 months after the last study enrollment. All study required visits will be completed as part of regularly scheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or above, or above legal age to give informed consent specific to state and national law
2. Willing and capable of providing informed consent
3. Planned to be implanted or replaced with a VISIONIST Ingenio 2 CRT-P device
4. Planned to be implanted with a 3-lead CRT-P system
5. Planned to be connected to the remote data collection through the Latitude® system
6. Able to do a 6 minute walk test
7. Maximum sensor rate of age predicted maximal heart rate (APMHR) 80% should be clinically acceptable
8. Willing and capable of participating in all visits associated with this study at an approved clinical study center and at the intervals defined-

Exclusion Criteria:

1. Documented life expectancy of less than 12 months
2. Currently on the active heart transplant list
3. Enrolled in any other concurrent study without prior written approval from Boston Scientific, with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict and do not affect the following:

   * Schedule of procedures for the Rally CRT-P Study (i.e., should not cause additional or missed visits)
   * Rally CRT-P Study outcomes (i.e., involve medications that could affect the heart rate of the subject)
   * Conduct of the Rally CRT-P Study per Good Clinical Practice (GCP)/ International Standard Organization (ISO) 14155:2011/ local regulations as applicable
4. In chronic atrial fibrillation
5. APMHR needs to be programmed < 80%.
6. Not planned to receive a functional atrial lead
7. Per the implanting physician's discretion, subject is not a suitable candidate to receive the study device as determined during the implant procedure
8. Women of childbearing potential who are or might be pregnant at the time of study enrollment
9. Unwilling or unable to participate in all scheduled study follow up visits at an approved study center
10. Does not anticipate being a resident of the area for the scheduled duration of the trial. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned to be implanted or replaced with a VISIONIST Ingenio 2 CRT-P device
  The Ingenio 2 CRT-Ps are indicated for patients who have symptomatic congestive heart failure (CHF) including left ventricular (LV) dysfunction and wide QRS, and/or one or more of the following conditions:
  Symptomatic paroxysmal or permanent second- or third-degree atrioventricular (AV) block Symptomatic bilateral bundle branch block Symptomatic paroxysmal or transient sinus node dysfunction with or without associated AV conduction disorders (i.e., sinus bradycardia, sinus arrest, sinoatrial [SA] block) Bradycardia-tachycardia syndrome, to prevent symptomatic bradycardia or some forms of symptomatic tachyarrhythmias Neurovascular (vaso-vagal) syndromes or hypersensitive carotid sinus syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Pakarinen, Dr., Principal Investigator — Helsinki University Central Hospital
Locations (8):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Germany (6):
  - Unfallkrankenhaus Berlin, Berlin
  - Herz-und Gefäßzentrum Göttingen, Göttingen
  - Krankenhaus Landshut-Achdorf, Landshut
  - University Magdeburg, Magdeburg
  - Klinikum Oldenburg, Oldenburg
  - Harzklinikum Quedlinburg, Quedlinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 11 May 2015 and the study was completed on 22 March 2017, which corresponds to the last visit of the last subject. A total of 64 subjects across 8 centers were enrolled in Finland and Germany.
Groups:
- Actively Enrolled Patients: Patients actively enrolled and implanted with a 3-lead CRT-P system.
Period: Overall Study
Arm/Group | Actively Enrolled Patients
Started | 64
Completed | 54
Not Completed | 10
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Consent ineligible | 1
Not completed — Did not undergo implant procedure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Actively Enrolled Patients
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 15
  Germany | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without CRT-P Device Related Complications
Description: Evaluate the Device-Related Complication Free Rate (DRCFR) at 3 months post-implant, which was based on complications that were related to the CRT-P device. A device-related complication was an adverse event that resulted in death, serious injury, a correction using invasive intervention or permanent loss of device functions, and that was assessed as related to the device.
Time Frame: 3 months post-implant
Population: Out of 61 actively enrolled subjects (3 subjects were not implanted with the study device), 55 patients continued the study for at least 3 months: 6 subjects were excluded from analysis because either they died or withdrew before 3 months analysis, or because no 3 months data was available.
Measure: Number (90% Confidence Interval); unit: % of participants
Groups:
- Actively Enrolled Patients: Subjects actively enrolled and implanted with a 3-lead CRT-P system.
Arm/Group | Actively Enrolled Patients
Number analyzed (Participants) | 55
% of participants | 100 [94.7 to 100]
Statistical Analysis 1: Comparison: Actively Enrolled Patients; Test type: Other; p < 0.001, exact binomial rate

2. Primary Outcome: LV Pacing Threshold
Description: Primary Effectiveness endpoint: evaluation of the left ventricular pacing threshold measurements performed at 0.5 ms pulse width at 3 months post-implant.
Time Frame: 3 months post-implant
Population: 61 actively enrolled subjects were included in the analysis. 3 subjects did not receive the study device.
Measure: Mean (90% Confidence Interval); unit: Volt
Arm/Group | Actively Enrolled Patients
Number analyzed (Participants) | 61
Volt | 1.65 [1.38 to 1.93]
Statistical Analysis 1: Comparison: Actively Enrolled Patients; Test type: Other; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events are collected from enrollment throughout study completion (last subject last visit)
Description: All adverse events are collected as per ISO 14155:2011 and medical device guidance (MEDDEV) 2.7/3 12/2010
Arm/Group | Actively Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 3/61
Serious Adverse Events (participants affected / at risk) | 20/61
Other Adverse Events (participants affected / at risk) | 40/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Actively Enrolled Patients (N=61)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Other SVT (Cardiac disorders) | 1 (1)
Renal (Renal and urinary disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Coronary Artery Disease (Vascular disorders) | 1 (1)
Pulmonary edema - heart failure (Cardiac disorders) | 1 (1)
Heart failure symptoms - unspecified (Cardiac disorders) | 1 (1)
Chest pain - ischemic (Cardiac disorders) | 1 (1)
Dyspnea (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
LV - elevated threshold (Product Issues) | 1 (1)
LV - extracardiac stimulation (Product Issues) | 1 (1)
Procedure - coronary venous dissection (Surgical and medical procedures) | 1 (1)
RA - dislogement - elevated threshold (Product Issues) | 1 (1)
RV - dislodgement - elevated threshold (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Actively Enrolled Patients (N=61)
Atrial Fibrillation (Cardiac disorders) | 4 (6)
Device Deficiency (Product Issues) | 2 (2)
Dyspnea - Heart failure (Cardiac disorders) | 1 (1)
Elevated threshold - RA (Product Issues) | 1 (1)
Extracardiac stimulation - LV (Product Issues) | 3 (4)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Hematoma - Pocket (<= 30 days post-implant) (Surgical and medical procedures) | 1 (1)
Inability to maintain telemetry (Product Issues) | 1 (1)
Infection (> 30 days post-implant) (Product Issues) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2)
Other - Lead - Procedure (Product Issues) | 2 (2)
Other- Patient condition - Cardiovascular (Cardiac disorders) | 1 (1)
Other- Patient condition - Non- cardiovascular (General disorders) | 1 (1)
Pacemaker-mediated tachycardia (PMT) (Product Issues) | 10 (16)
Pneumothorax - Procedure (Surgical and medical procedures) | 1 (1)
Post-surgical wound discomfort (Surgical and medical procedures) | 1 (1)
Premature atrial contractions (PAC) (Cardiac disorders) | 1 (1)
Premature ventricular contractions (PVC) (Cardiac disorders) | 6 (11)
Syncope (Cardiac disorders) | 1 (1)
Undersensing - RA (Product Issues) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT02488239/Prot_SAP_000.pdf